CLINICAL TRIAL: NCT02726360
Title: Physician Use of Non-English Language Skills in Cancer Care
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Edward-Elmhurst Health System (Other); Johns Hopkins University (Other); Lincoln Medical and Mental Health Center (Other); Queens Cancer Center of Queens Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-316
Record Dates: First submitted 2016-03-15; First posted 2016-04-01 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Colon Cancer; Lung Cancer
Keywords: Communication; 15-316; Physician; Use; Non-English; Language Skills
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Communication | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Oncology physician: Physicians (MD or DO) in the oncology departments of participating hospitals will complete a survey. Non-English language proficiency will be assessed by self-assessment using Interagency Language Roundtable (ILR) scale, which the PI has previously used. The physician survey is collected among treating physicians of patients enrolled to MSK IRB approved protocols 12-099 and 12-223 at some of the participating hospitals. For physicians who already completed this survey as part of participation in protocol 12-099 or 12-223, data will be extracted from the respective study's REDCap database.
  Interventions: Behavioral: survey; Behavioral: Audio record
- patients: Audio record the initial visits between patients and their treating physician. Analyze 48 patient-physician dyad recordings using the Roter Interaction Analysis System (RIAS).
  Interventions: Behavioral: Audio record

INTERVENTIONS:
Behavioral: survey — The ILR Scale, a non-English language proficiency self-assessment.
  Other Names: ILR Scale
  Groups: Oncology physician
Behavioral: Audio record — Audio record the initial visits between patients and their treating physician

SUMMARY:
The purpose of this study is to test a method for analyzing interactions between patients and doctors, the Roter Interaction Analysis System (RIAS). The RIAS measures the quality of communication between patients and their cancer doctors.

ELIGIBILITY:
Inclusion Criteria:

* is a English or Spanish-speaking patient
* between the ages of 21-80 years old
* has a new diagnosis of any type of cancer (diagnosed within the past 4 months), or has a recurrence of either breast, colon or lung cancer (recurrence diagnosed within the past 4 months)
* scheduled to have surgery or begin chemotherapy and/or radiation therapy within the next 2 months

Oncology clinician Inclusion:

* provides care to LEP patients
* has MD, DO, RN, NP or PA degree
* is between the ages of 21-80

Exclusion Criteria:

* is unable to provide informed consent in either English or Spanish

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll all treating physicians of participating sites who are likely to treat LEP Spanish-speaking patients. All patient recruitment will be done by bilingual research staff who are consenting professionals with (when necessary) a volunteer affiliation with the collaborating study site.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
study-specific coding structure | 2 years
  using the RIAS in cancer care across English and Spanish languages will be assessed by evaluating whether this existing, validated coding system 'works' across a language barrier.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Diamond, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Elmhurst Hospital Center, Queens, New York
  - Lincoln Medical Center, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT02726360/ICF_000.pdf